CLINICAL TRIAL: NCT05917899
Title: Virtual Family-Centered Rounds for Caregivers With Limited English Proficiency: A Feasibility Trial
Brief Title: Limited English Proficiency Virtual Family-Centered Rounds
Acronym: LEP vFCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1736147
Record Dates: First submitted 2023-06-06; First posted 2023-06-26 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Pediatric Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Family-Centered Rounds (Experimental): Parents/guardians of the hospitalized infants will be invited to join family-centered rounds virtually plus usual care (usual care is the ability to join family-centered rounds in person or not to join at all).
  Interventions: Behavioral: Virtual Family-Centered Rounds

INTERVENTIONS:
Behavioral: Virtual Family-Centered Rounds — The care team will use a computer with a speaker camera, mounted on a stand with wheels to launch telehealth visits using the application ExtendedCare. This platform meets HIPAA security rules and launches from the patient's electronic health record. From within this telehealth visit, a care team member will send a message (via text or email) to the parent(s) that includes a link that can be clicked to open a browser that allows the parent to join the telehealth visit. Parent do not need to download or use an application. The care team will invite the video interpreter to join the visit if a parent is present. Family-centered rounds will then proceed in usual fashion with the care team and [if in attendance] parent(s). Parents can participate in virtual family-centered rounds as much, or as little, as they choose.

SUMMARY:
This study will be a pilot test of using telehealth with an interpreter as an additional option for parents with limited English proficiency to join family-centered rounds in the neonatal intensive care unit.

ELIGIBILITY:
We will enroll family units. Family units consist of the hospitalized infant and their eligible parents/guardians.

Inclusion Criteria - INFANT:

* Infants aged less than 365 days who are admitted to the neonatal intensive care unit
* Have at least one eligible parent or guardian (see below for parent eligibility criteria)

Exclusion Criteria - INFANT:

* Have restrictions placed by child protective services, including visitation restrictions or restricted access to patient information
* Infants with a previous neonatal intensive care unit admission (and enrollment) during the trial period
* Infants already enrolled in a different trial that includes a virtual family-centered rounds intervention

Inclusion Criteria - PARENT:

* Aged 18 years or older
* Preferred language that is other than English
* Have at least one infant enrolled in the trial

Exclusion Criteria - PARENT:

* Under age 18 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Family-Centered Rounds Parent Attendance | From date of randomization until the date of disposition from the neonatal intensive care unit for any cause (assessed up to 396 days)
  Proportion of the number of weekday round encounters with at least one parent present - either virtually or in-person - divided by the infant's total number of weekday round encounters

SECONDARY OUTCOMES:
Patient length of stay | From date of admission to the neonatal intensive care unit until the date of disposition from the unit for any cause (assessed up to 396 days)
  Days in the neonatal intensive care unit. Obtained from electronic health record.
Breastmilk feeding at discharge | Date of disposition from the neonatal intensive care unit for any cause (assessed up to 396 days)
  Dichotomous outcomes. Include (a) breastmilk feeding initiation, (b) any breastmilk feeding at the time of discharge from the neonatal intensive care unit, and (c) exclusive breastmilk feeding at the time of discharge from the neonatal intensive care unit. Breastmilk feeding includes consuming milk from the birth parent via any delivery method (e.g., bottle, feeding tube, breast). Any breastmilk feeding will be defined as the infant consuming any amount of milk from the birth parent, with or without the addition of formula or fortifier. Exclusive breastmilk feeding will be defined as 100% of base feeding type as milk from the birth parent, with or without a bovine or human fortifier. Obtained from electronic health record (0 days)
Medical errors and adverse events | Date of disposition from the neonatal intensive care unit for any cause (assessed up to 396 days)
  Include the rates of harmful errors, non-harmful errors, and overall errors (harmful errors plus non-harmful errors). Obtained via review of data from electronic health record and solicited reports. Two neonatologists will independently categorize each event as a harmful error (preventable adverse event), non-harmful error, non-preventable adverse event, or exclusion.
Patient Experience | Date of disposition from the neonatal intensive care unit for any cause (assessed up to 396 days)
  Unit of measure: mean score; Measure/Tool: Emergency Department CAHPS (Consumer Assessment of Healthcare Providers and Systems) (parent survey, 2 items measuring overall experience).
Patient Activation | Date of disposition from the neonatal intensive care unit for any cause (assessed up to 396 days)
  Unit of measure: mean score; Measure/Tool: Parent-Patient Activation Measure (P-PAM) (parent survey)
Parent Quality of Life | Date of disposition from the neonatal intensive care unit for any cause (assessed up to 396 days)
  Unit of measure: mean score. Measure/Tool: PedsQL Family Impact Module (parent survey)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoyt-Austin AE, Zerda EN, Tancredi DJ, Marcin JP, Ketchersid A, Horath ET, Bushong TR, Merriott DS, Romano PS, Hoffman KR, Rosenthal JL. Protocol for a single-arm feasibility trial of virtual family-centered rounds: increasing opportunities for family engagement among caregivers with language preference other than English. Pilot Feasibility Stud. 2025 Feb 12;11(1):16. doi: 10.1186/s40814-025-01599-4. PMID 39940014